CLINICAL TRIAL: NCT05175209
Title: The Effect of Ulnar Nerve Entrapment Localization on Ipsilateral Upper Extremity Functions in Patients With Ulnar Nerve Entrapment Neuropathy.
Brief Title: The Effect of Ulnar Nerve Entrapment Localization on Ipsilateral Upper Extremity Functions. The Effect of Ulnar Nerve Entrapment Localization on Ipsilateral Upper Extremity Functions. The Effect of Ulnar Nerve Entrapment Localization on Ipsilateral Upper Extremity Functions.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Volkan Şah, Principal Investigator., Yuzuncu Yil University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Hundredth Year University
Record Dates: First submitted 2021-12-13; First posted 2022-01-03 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Ulnar Neuropathies
MeSH Terms: conditions — Ulnar Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electromyelography (Other): EMG will be performed only once to determine the ulnar nerve entrapment site in patients.
  Interventions: Diagnostic Test: EMG

INTERVENTIONS:
Diagnostic Test: EMG — Electromyelography

SUMMARY:
Regardless of the cause of ulnar nerve entrapment neuropathy, investigators are planning to explore the relationship between the ipsilateral upper extremity dysfunction that may develop due to ulnar neuropathy and the level of entrapment in electromyelography.

ELIGIBILITY:
Inclusion Criteria:

* having ulnar nerve entrapment neuropathy with clinical examination and EMG (electroneuromyography)
* to be between the ages of 18-65
* be give informed consent

Exclusion Criteria:

* inflammatory arthritis
* hemiplegia
* contractures of shoulder-arm-hand joints

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-03-20 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Disabilities of the Arm, Shoulder and Hand (DASH) score | 10 minutes.
  Evaluation of upper extremity function between 0 and 100 points, higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No